CLINICAL TRIAL: NCT00033241
Title: A Phase Ib Multicenter Trial To Determine The Safety, Tolerance And Preliminary Antineoplastic Activity Of Gemcitabine Administered In Combination With Escalating Oral Doses Of OSI-774 To Patient Cohorts With Recently Diagnosed, Gemcitabine-Naive, Advanced Pancreatic Carcinoma Or Other Potentially Responsive Malignancies
Brief Title: Erlotinib Combined With Gemcitabine in Treating Patients With Newly Diagnosed Locally Advanced or Metastatic Pancreatic Cancer or Other Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OSI Pharmaceuticals (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Purpose: Treatment
Other Study IDs: OSI-774-155; CDR0000069266; UARIZ-HSC-01128; NCI-V02-1694
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2015-06

CONDITIONS: Pancreatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; unspecified adult solid tumor, protocol specific; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride; Gemcitabine

INTERVENTIONS:
Drug: erlotinib hydrochloride
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Erlotinib may interfere with the growth of tumor cells and slow the growth of the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining erlotinib with gemcitabine may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining erlotinib with gemcitabine in treating patients who have newly diagnosed locally advanced or metastatic pancreatic cancer or other solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of erlotinib in combination with gemcitabine in patients with recently diagnosed, gemcitabine-naive, locally advanced or metastatic pancreatic carcinoma or other potentially responsive solid tumor.
* Determine the safety and tolerability of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine the objective antitumor response rate and response duration in patients treated with this regimen.
* Determine the time to disease progression and duration of overall survival in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of erlotinib.

Patients receive gemcitabine IV over 30 minutes on day 1 of weeks 1-7 and oral erlotinib once daily beginning on day 3 of week 1 and continuing for 8 weeks (course 1). Patients receive subsequent courses of therapy comprising gemcitabine once weekly for 3 weeks and erlotinib once daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 12 additional patients are accrued and treated at the MTD as above.

Patients are followed at 30 days.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study within 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed locally advanced or metastatic epithelial carcinoma of the pancreas or other malignancy considered to be potentially responsive to gemcitabine

  * Newly diagnosed or gemcitabine naive
* Measurable or evaluable disease
* Not amenable to surgical intervention due to medical contraindications or non-resectability of the tumor
* No islet cell tumors or other non-epithelial cell carcinomas of the pancreas
* No active CNS metastases or leptomeningeal disease

  * Treated or asymptomatic brain metastases are allowed if on a stable dose of corticosteroids and/or there is no change in brain disease status for at least 4 weeks after related therapy (e.g., whole-brain radiotherapy)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL (except for documented Gilbert's syndrome)
* AST or ALT less than 2 times upper limit of normal (ULN) (no greater than 5 times ULN if hepatic obstruction or metastases present)
* Albumin at least 2.5 g/dL

Renal:

* Creatinine less than 1.5 times ULN OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No significant cardiovascular disease
* No history of congestive heart failure currently requiring therapy
* No ventricular arrhythmia requiring anti-arrhythmic therapy
* No severe conduction disturbances
* No angina pectoris requiring therapy
* No myocardial infarction within the past 6 months

Gastrointestinal:

* No significant gastrointestinal abnormalities including:

  * Requirement for IV alimentation
  * Active peptic ulcer disease

Ophthalmic:

* No significant ophthalmologic abnormalities including:

  * Severe dry eye syndrome
  * Keratoconjunctivitis sicca
  * Sjogren's syndrome
  * Severe exposure keratopathy
  * Disorders that would increase the risk for epithelium-related complications (e.g., bullous keratopathy, aniridia, severe chemical burns, or neutrophilic keratitis)
  * Abnormal Schirmer test (less than 2 mm) allowed provided there is no evidence of clinically significant corneal surface abnormalities

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known or suspected hypersensitivity to gemcitabine
* No uncontrolled infection
* HIV negative
* No other malignancy within the past 5 years except treated non-melanoma skin cancer or carcinoma in situ of the breast or cervix
* No other life-threatening illness
* No psychiatric disorders or altered mental status the would preclude informed consent or study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 28 days since prior immunotherapy or biological response modified therapy for the primary malignancy
* No concurrent immunotherapy or biologic response modifier therapy for the primary malignancy

Chemotherapy:

* See Disease Characteristics
* At least 28 days since prior chemotherapy for the primary malignancy
* No prior mitomycin or nitrosoureas for the primary malignancy
* No more than 6 prior courses of chemotherapy with an alkylating agent for the primary malignancy
* No prior gemcitabine for the primary malignancy except as a low-dose (less than 500 mg/m^2) radiosensitizer administered concurrently with or within 2 weeks after radiotherapy at least 3 months ago
* No other concurrent chemotherapy for the primary malignancy

Endocrine therapy:

* See Disease Characteristics
* At least 28 days since prior systemic hormonal therapy (except LH-RH agonists) for the primary malignancy
* No concurrent systemic hormonal therapy (except LH-RH agonists) for the primary malignancy
* Other concurrent endocrine therapy is allowed as follows:

  * Hormonal therapy (e.g., megestrol) for appetite stimulation
  * Nasal, ophthalmic, or topical glucocorticoids
  * Oral glucocorticoids for adrenal insufficiency
  * Low-dose maintenance steroids

Radiotherapy:

* See Disease Characteristics
* At least 28 days since prior radiotherapy for the primary malignancy or metastases and recovered
* No prior wide-field radiotherapy to 25% or more of marrow-bearing bone
* No prior pelvic irradiation
* No concurrent radiotherapy for the primary malignancy or metastases
* No concurrent wide-field radiotherapy for pain management

Surgery:

* See Disease Characteristics
* Recovered from any prior surgery
* No prior surgical procedures affecting absorption

Other:

* No prior agent for the primary malignancy targeting the epidermal growth factor receptor (EGFR) or EGFR-specific tyrosine kinase activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-07-23 (Actual); Primary Completion 2004-04-22 (Actual); Study Completion 2004-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Santabarbara, MD, Study Chair — OSI Pharmaceuticals
Locations (2):
- United States (2):
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Cancer Therapy and Research Center, San Antonio, Texas

REFERENCES:
- [Result] Dragovich T, Patnaik A, Rowinsky EK, et al.: A phase I B trial of gemcitabine and erlotinib HCL in patients with advanced pancreatic adenocarcinoma and other potentially responsive malignancies. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-895, 2003.
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=61